CLINICAL TRIAL: NCT02215798
Title: Post-Marketing Surveillance Study on the Safety and Efficacy of Cymbalta (Duloxetine) on Diabetic Peripheral Neuropathic Pain Among Filipino Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1208.31
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cymbalta
  Interventions: Drug: Cymbalta

INTERVENTIONS:
Drug: Cymbalta

SUMMARY:
Primary objective: To estimate the frequency of adverse events, serious and non-serious in Filipino patients with diabetic peripheral neuropathic pain treated with duloxetine 60mg once daily within the study duration of approximately 6-8 weeks in a naturalistic clinical setting. Secondary objective: To evaluate the change from baseline to endpoint in the Brief Pain Inventory (BPI) and Neuropathic Pain Questionnaire (NPQ) assessed by the investigators in duloxetine use in the treatment of diabetic peripheral neuropathic pain among Filipino patients within the study duration of approximately 6-8 weeks in a naturalistic clinical setting.

ELIGIBILITY:
Inclusion Criteria

* Are of Filipino race
* Are male or female outpatients at least 18 years of age
* Provide written consent to the release of their data after being informed of the study
* Are known diabetics and have been clinically diagnosed by the investigator to have Diabetic Peripheral Neuropathic Pain
* Are judged by the investigator to be reliable, and agree to keep appointments for clinic visits, complete tests and procedures as may be required by his/her attending physician in the course of routine clinical care
* Treated with duloxetine according to the approved Product Information as prescribed by the investigator in the routine care of the patient, without the concomitant conditions and medications specified therein as contraindicated

Exclusion criteria

* Are the investigators or their immediate families. Immediate family was defined as the investigator's spouse, parents, naturally or legally adopted child (including stepchild living in the investigator's household), grandparents, or grandchild. Employees of investigators are also not eligible
* Are simultaneously participating in a different study that includes a treatment intervention and/or an investigational drug
* Are hypersensitive to duloxetine or any of its components
* Are pregnant and/or nursing mothers
* Have concomitant conditions contraindicated for duloxetine treatment, as described in the Product Information (e.g. liver disease resulting in hepatic impairment, severe renal impairment)
* Are concomitantly taking contraindicated medications, as described in the Product Information (e.g. fluvoxamine, ciprofloxacin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2006-07; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Frequency of serious and non-serious adverse events | up to 8 weeks

SECONDARY OUTCOMES:
Change from baseline in Brief Pain Inventory (BPI) | up to 8 weeks
Change from baseline in Neuropathic Pain Questionnaire (NPQ) | up to 8 weeks